CLINICAL TRIAL: NCT02357316
Title: Heritability and Genetics of Fat Taste
Status: Completed | Type: Observational
Sponsor: Purdue University (Other)
Collaborators: Denver Museum of Nature & Science (Unknown)
Responsible Party: Principal Investigator, Richard Mattes, dir of public health/dist prof nutr sc, Purdue University
Other Study IDs: 055-039
Record Dates: First submitted 2014-11-20; First posted 2015-02-06 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Healthy
Keywords: Taste responses of healthy individuals

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Buccal cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All participants: All individuals visiting the museum who want to participate and sign a consent form.

SUMMARY:
The investigators seek to determine how genetics and the environment influence the ability to taste and smell fat. The investigators believe that people who consume higher fat diets and people who have higher body fat levels are less able to taste and smell fat. The investigators expect to see that people who are less able to taste and smell fat will share certain genetic differences.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate
* Ages 8 and older

Exclusion Criteria:

* Younger than 8 years old

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy individuals ages 8 and older
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2013-11 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Taste sensitivity | At visit
  Intensity ratings of linoleic acid will be measured using a visual analog scale.
Genotype | At visit
  Various SNPs related to taste will be genotyped.
Anthropometric measures | At visit
  BMI, % body fat, % body water will be measured using BIA.
Dietary data | At visit
  Exposure to high-fat foods and information from most recent meal (optional) will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Denver Museum of Nature & Science, Denver, Colorado, United States